CLINICAL TRIAL: NCT05347134
Title: A Randomized, Controlled, Open-label, Multi-center Phase III Clinical Trial of SKB264 for Injection Versus Investigator Selected Regimens in Patients With Unresectable Locally Advanced, Recurrent or Metastatic Triple-negative Breast Cancer Who Have Failed Second-line or Above Prior Standard of Care
Brief Title: SKB264 Injection vs Investigator Selected Regimens to Treat Locally Advanced, Recurrent or Metastatic Triple-negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅲ-03
Record Dates: First submitted 2022-04-15; First posted 2022-04-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — eribulin; Capecitabine; Gemcitabine; Vinorelbine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into the experiment group and control group in a 1:1 ratio, stratified by: number of previous treatment lines (2-3 vs. >3); Presence of liver metastases (yes vs. No)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKB264 (Active Comparator): 5 mg/kg, IV (in the vein) on day 1 and Day 15 of each 28 day cycle.
  Interventions: Drug: SKB264
- Eribulin or Capecitabine or Gemcitabine or Vinorelbine (Active Comparator): Eribulin:1.4mg/m2, IV (in the vein) on day 1 and Day 8 of each 21 day cycle.
  Capecitabine:1000-1250mg/m2, po,bid, from day 1 to Day 15 of each 21 day cycle.
  Gemcitabine:800-1000 mg/m2, IV (in the vein) on day 1 and Day 8 of each 21day cycle.
  Vinorelbine:25 mg/m2, IV (in the vein) on day 1 and Day 8 of each 21 day cycle.
  Interventions: Drug: SKB264

INTERVENTIONS:
Drug: SKB264 — SKB264 ：5 mg/kg, IV (in the vein) on day 1 and Day 15 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Eribulin:1.4mg/m2, IV (in the vein) on day 1 and Day 8 of each 281day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Capecitabine:1000-1250mg/m2, po,bid, from day 1 to Day 15 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Gemcitabine:800-1000 mg/m2, IV (in the vein) on day 1 and Day 8 of each 281day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Vinorelbine:25 mg/m2, IV (in the vein) on day 1 and Day 8 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Eribulin; Capecitabine; Gemcitabine; Vinorelbine

SUMMARY:
The purpose of this study is to evaluate the efficacy of SKB264 in patients with unresectable locally advanced, recurrent or metastatic triple-negative breast cancer who have failed second-line or above prior standard of care

DETAILED DESCRIPTION:
The 2021 CSCO guidelines recommend treatment for patients with advanced TNBC as follows: Taxoides are generally preferred for patients who have failed anthracycline therapy in the past; For patients with anthracycline and taxane treatment failure, there is no standard therapy. Previously unused chemotherapy alone or in combination can be considered. However, the toxicity of combination chemotherapy is high and the survival benefit is limited, therefore, in consideration of the quality of life of advanced patients, single-agent chemotherapy is recommended as a priority.

ELIGIBILITY:
Inclusion Criteria:

Subjects will not be included unless they meet all of the following criteria:

1. Males or females age 18 to 75 years old (inclusive) at the time of signing the informed consent form;
2. Histologically and/or cytologically confirmed TNBC based on pathology reports on recent biopsy specimens or other pathological samples (central laboratory confirmation is not required), including:

   1. Definition of human epidermal growth factor receptor 2 (HER2) negative: immunohistochemistry (IHC) of 0 or 1+; if HER is 2+ by IHC, negative HER2 expression must be confirmed by fluorescence in situ hybridization (FISH).
   2. Estrogen and progesterone receptor negative means that less than 1% of the cells express hormone receptors as indicated by IHC;
3. Patients with unresectable locally advanced or metastatic triple-negative breast cancer who have received at least two lines of standard of care regimens, including:

   1. Any treatment received by the patients regardless of triple-negative state can be included as one of the standard of care regimens;
   2. For patients whose treatment regimens have been changed due to intolerability to toxicity, the intolerable regimens can be included as one of the prior standard of care regimens;
   3. For neoadjuvant and/or adjuvant chemotherapy, if relapse or disease progression to unresectable locally advanced or metastatic disease occurs during treatment or within 12 months after discontinuation of treatment (at least 2 cycles have been completed), it will be considered as one of the standard of care regimens. And the patients must also have received one therapy and have progressed on this therapy during the stage of unresectable locally advanced or metastatic disease;
   4. For patients with documented germline BRCA1/BRCA2 mutations, if they have been treated with an approved PARP inhibitor, then the PARP inhibitor can be considered as one of the 2 prior standard of care regimens required;
   5. Patients must have progressed on or were intolerable to the treatment during or after the last treatment prior to enrollment;
4. All patients must have been previously treated with taxanes; and those who have been treated with taxanes for at least 1 cycle and show contraindications or intolerability during or at the end of the cycle can be included, regardless of the disease stage during this treatment;
5. Patients must have at least one measurable lesion per RECIST v1.1 criteria; those with only skin or bone lesions cannot be included;
6. Subjects with a Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 with an expected survival of ≥ 12 weeks;
7. Subjects must provide tumor tissues or tissue specimens;
8. Subjects must have adequate organ and bone marrow function (no blood transfusion, recombinant human thrombopoietin, or colony stimulating factor therapy has been received within 2 weeks prior to the screening), which is defined as follows:

   1. Hematology: neutrophil count (NEUT) ≥ 1.5 × 109 /L; platelets (PLT) ≥ 100 × 109 /L; hemoglobin ≥ 9 g/dL;
   2. Liver function: aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 × upper limit of normal (ULN); total bilirubin (TBIL) ≤ 1.5 × ULN; for patients with liver metastases, ALT and AST must be ≤ 5 × ULN, TBIL ≤ 2 × ULN; for patients with liver or bone metastases, ALP must be ≤ 5 × ULN;
   3. Albumin ≥ 3 g/dL;
   4. Renal function: creatinine clearance (Ccr) ≥ 60 ml/min (see Annex for Cockcroft-Gault formula);
   5. Coagulation function: international normalized ratio (INR), activated partial thromboplastin time (APTT) and prothrombin time (PT) ≤ 1.5 × ULN;
9. Subjects must have recovered from all toxicities (except alopecia) due to prior treatments to ≤ grade 1 based on the assessment per CTCAE 5.0 criteria;
10. Subjects voluntarily participate in the study, sign the informed consent form, and will be able to comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded:

1. Patients with a history of central nervous system (CNS) metastases or current CNS metastases;
2. Patients with other malignancies, except cured basal or squamous cell skin cancer or in situ cancer of cervix; and patients with other malignancies must have a tumor-free period of at least 5 years;
3. Patients with Gilbert's disease;
4. Patients who have received prior TROP2-targeted therapy;
5. Patients who have received live vaccines within 30 days prior to the first dose;
6. Patients who required the treatment of strong inhibitors or inducers of cytochrome P450 3A4 enzyme (CYP3A4) within 2 weeks prior to the first dose and during the study treatment (strong inhibitors or inducers of CYP3A4 are not allowed in this study, and representative drugs of strong CYP3A4 inhibitors or inducers are listed in the Annex). Patients who received continued high dose of systemic corticosteroids within 2 weeks prior to the first dose (low-dose corticosteroids, such as ≤ 10 mg daily prednisone or equivalent, are allowed if the dose is stable for 4 weeks);
7. Patients who have received any chemotherapy, hormonal therapy, radiotherapy, immunotherapy, biological therapy or other drugs within 4 weeks prior to the first dose of study treatment or within 5 half-lives of the drug used in the previous period (whichever is shorter), or received treatment with traditional Chinese medicine preparations for approved anti-tumor indications 2 weeks prior to the first dose of study treatment, or received major surgeries 4 weeks prior to the first dose of study treatment;
8. With concomitant infections requiring systemic antibiotic therapy within 1 week prior to the first dose of study treatment;
9. Presence of any serious and/or uncontrolled comorbidities that prevent the patient from participating in the study, such as:

   1. Impaired cardiac function, including any of the following: (not necessarily all of the following):

      aa) Corrected QT interval (QTcF) between ventricular depolarization to repolarization > 480 ms at baseline; ab) Left ventricular ejection fraction (LVEF) < 50% as indicated by echocardiography (ECHO) ;
   2. Other clinically significant heart diseases, including any of the following known medical history:

      ba) Angina pectoris; bb) Congestive cardiac failure; bc) Myocardial infarction;
   3. Patients with (noninfectious) interstitial lung disease (ILD) or history of pneumonia requiring steroid therapy; patients with serious pulmonary function impairment due to lung disease;
   4. Patients with current or previous active chronic inflammatory bowel disease or intestinal obstruction or gastrointestinal (GI) perforation;
   5. Uncontrolled hypertension (systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg), with a history of unstable hypertension, or with a history of poor compliance with antihypertensive treatment;
   6. Uncontrolled diabetes (fasting glucose ≥ 10 mmol/L and/or glycated hemoglobin (HbA1c) ≥ 8%);
10. Active hepatitis B (hepatitis B surface antigen positive, and HBV-DNA above 500 IU/ml or 1x ULN, whichever is higher) or hepatitis C (hepatitis C antibody positive, and HCV-RNA above 1x ULN); with known history of positive human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS); positive syphilis antibody test;
11. History of serious drug allergy, with known allergy to macromolecular protein preparations or any component of the study drug formulation;
12. Pregnant or lactating women; or patients of childbearing potential (male or female) who cannot use effective medical contraception during the study treatment period and for 6 months after the end of the dosing period (see Annex for specific contraceptive measures);
13. During the screening process prior to the first dose, the condition deteriorated rapidly, such as severe changes in performance status, unstable pain requiring adjustment of analgesic therapy;
14. Other circumstances that, in the opinion of the investigator, are not appropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  Progression-free survival (PFS) as assessed by an Independent Review Committee (IRC) based on RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival(PFS) | up to 24 months
  Progression-free survival (PFS) assessed by the investigators according to RECIST V 1.1
Objective Response Rate (ORR) | up to 24 months
  The percentage of patients with CR and PR assessed by the Independent Review Committee and investigators according to RECIST v 1.1
Disease Control Rate (DCR) | up to 24 months
  The proportion of patients who have achieved CR，PR and SD assessed by the Independent Review Committee and investigators according to RECIST v 1.1
Duration of Response (DoR) | up to 24 months
  From the date that response criteria are first met to the first occurrence of PD as determined by the Independent Review Committee and investigators according to RECIST v1.1 or death from any cause, whichever occurs first
Overall Survival (OS) | up to 24 months
  OS, defined as the time from randomization to death or lose of follow, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Jiangsu Province Hospital, Nanjing, Jiangsu

REFERENCES:
- [Derived] Yin Y, Fan Y, Ouyang Q, Song L, Wang X, Li W, Li M, Yan X, Wang S, Sun T, Teng Y, Tang X, Tong Z, Sun Z, Ge J, Jin X, Diao Y, Liu G, Xu B. Sacituzumab tirumotecan in previously treated metastatic triple-negative breast cancer: a randomized phase 3 trial. Nat Med. 2025 Jun;31(6):1969-1975. doi: 10.1038/s41591-025-03630-w. Epub 2025 Apr 11. PMID 40217078